CLINICAL TRIAL: NCT00912925
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Multinational, Clinical Study of Recombinant Human Alpha L-Iduronidase In Patients With Mucopolysaccharidosis I
Brief Title: Clinical Study of Aldurazyme in Patients With Mucopolysaccharidosis (MPS) I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: BioMarin/Genzyme LLC (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALID-003-99
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Results first posted 2009-08-19 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Mucopolysaccharidosis I; Hurlers Syndrome; Hurler-Scheie Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients in the placebo-control group were administered a solution of 100 millimolar (mM) sodium phosphate, 150 mM sodium chloride, and 0.001% polysorbate-80, adjusted to a pH of 5.8 administered intravenously over approximately 4 hours once weekly for 26 weeks.
  Interventions: Biological: Placebo
- Aldurazyme treatment (Active Comparator): Patients in the active treatment group received Aldurazyme intravenously at a dose of 100 Units/kg (approximately 0.58 mg/kg = labeled dose) administered intravenously over approximately 4 hours once weekly for 26 weeks.
  Interventions: Biological: rhIDU (recombinant human-Alpha-L-Iduronidase)

INTERVENTIONS:
Biological: rhIDU (recombinant human-Alpha-L-Iduronidase) — Patients in the active treatment group received Aldurazyme intravenously at a dose of 100 units/kg (approximately 0.58mg/kg) administered intravenously over approximately 4 hours once weekly for 26 weeks.
  Arms: Aldurazyme treatment
Biological: Placebo — Patients in the Placebo-control group were administered a solution of 100mM sodium phosphate , 150mM sodium chloride, and 0.001% polysorbate-80, adjusted to a pH of 5.8 administered intravenously over a time period of approximately 4 hours once weekly for 26 weeks.
  Arms: Placebo

SUMMARY:
This study is being conducted to demonstrate the safety and clinical efficacy of Aldurazyme treatment in MPS I patients

ELIGIBILITY:
Inclusion Criteria:

* The patient had a documented diagnosis of MPS I confirmed by measurable clinical signs and symptoms of MPS I and a fibroblast or leukocyte alpha-L-iduronidase enzyme activity level of less than 10% of the lower limit of the normal range of the measuring laboratory.
* Female patients of childbearing potential had a negative pregnancy test (urine-beta-human chorionic gonadotropin (hCG)) at baseline (all female patients of childbearing potential and sexually mature male patients were advised to use a medically accepted method of contraception throughout the study).
* The patient was capable of standing independently for 6 minutes and walking a minimum of 5 meters within 6 minutes.
* The patient was capable of performing a reproducible FVC maneuver.
* The patient had a baseline FVC value that was less than or equal to 80% of the patient's predicted normal FVC value based on polgar predicted values for standing height for children 5 through 7 years of age and the Hankinson predicted values for ages 8 and above.

Exclusion Criteria:

* The patient had undergone a tracheostomy.
* The patient had previously undergone a bone marrow transplantation.
* The patient was pregnant or lactating.
* The patient has received an investigational drug within 30 days prior to study enrollment.
* The patient had a medical condition, serious intercurrent illness, or other extenuating circumstance that could have significantly interfered with study compliance including all prescribing evaluations and follow-up activities.
* The patient had a known hypersensitivity to rhIDU or to components of the active or placebo test solutions.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2000-12; Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (4):
- United States (2):
  - New York, New York
  - Chapel Hill, North Carolina
- Vancouver, British Columbia, Canada
- Mainz, Germany

REFERENCES:
- [Derived] Tandon PK, Kakkis ED. The multi-domain responder index: a novel analysis tool to capture a broader assessment of clinical benefit in heterogeneous complex rare diseases. Orphanet J Rare Dis. 2021 Apr 19;16(1):183. doi: 10.1186/s13023-021-01805-5. PMID 33874971

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Aldurazyme Treatment
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Patients in the placebo-control group were administered a solution of 100 mM sodium phosphate, 150 mM sodium chloride, and 0.001% polysorbate-80, adjusted to a pH of 5.8 administered intravenously over approximately 4 hours once weekly for 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Aldurazyme Treatment | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Customized [Number; unit: participants]
  less than or equal to 12 years | 10 | 12 | 22
  13 to less than or equal to 18 years | 8 | 3 | 11
  19 to less than or equal to 65 years | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (7.63) | 15.6 (8.63) | 15.5 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 11 | 11 | 22
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 21 | 16 | 37
  Black | 0 | 0 | 0
  Hispanic | 0 | 4 | 4
  Asian | 1 | 1 | 2
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Change From Baseline to Week 26 in Percent Predicted Forced Vital Capacity (FVC)
Description: Percent Predicted Forced Vital Capacity (FVC): the maximal exhaled breathe volume following a maximal inhaled breath. Overall Change from Baseline to Week 26 in percent predicted FVC = (observed value)/(predicted value) * 100%). A higher value indicates a greater response.
Time Frame: Baseline to Week 26
Measure: Mean (Standard Deviation); unit: Percent predicted FVC
Arm/Group | Placebo | Aldurazyme Treatment
Number analyzed (Participants) | 23 | 22
Percent predicted FVC
  Baseline | 54.2 (16.00) | 48.4 (14.85)
  Week 26 | 51.5 (13.13) | 50.2 (17.10)
  Overall change from Baseline to Week 26 | -2.7 (7.12) | 1.8 (7.70)

2. Primary Outcome: Overall Change From Baseline to Week 26 in Six Minute Walk Test (6MWT)
Description: Six Minute Walk Test (6MWT): Distance walked (measured in meters) in 6 minutes. A longer distance indicates a greater response.
Time Frame: Baseline to Week 26
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | Aldurazyme Treatment
Number analyzed (Participants) | 23 | 22
meters
  Baseline | 366.7 (113.68) | 319.1 (131.41)
  Week 26 | 348.3 (128.82) | 338.8 (127.06)
  Overall change from Baseline to Week 26 | -18.4 (67.49) | 19.7 (68.56)

3. Secondary Outcome: Overall Change From Baseline to Week 26 in Apnea/Hypopnea Index (AHI)
Description: Apnea/Hypopnea Index (AHI): Number of absent (apnea) and shallow (hypopnea) breaths per hour of sleep. Overall change from Baseline to Week 26 in AHI. A greater decrease in events indicates a greater response.
Time Frame: Baseline to Week 26
Measure: Mean (Standard Deviation); unit: Events per hour
Arm/Group | Placebo | Aldurazyme Treatment
Number analyzed (Participants) | 19 | 20
Events per hour
  Baseline | 14.7 (15.20) | 20.5 (19.04)
  Week 26 | 15.5 (14.93) | 17.6 (16.75)
  Overall change from Baseline to Week 26 | 0.4 (8.55) | -2.9 (6.66)

4. Secondary Outcome: Overall Percent Change From Baseline to Week 26 in Liver Volume
Description: Liver Organ Volume: Volume of liver measured by Magnetic Resonance Imaging (MRI). Greater decrease in volume indicates a greater response.
Time Frame: Baseline to Week 26
Measure: Mean (Standard Deviation); unit: Cubic centimeters
Arm/Group | Placebo | Aldurazyme Treatment
Number analyzed (Participants) | 22 | 22
Cubic centimeters
  Baseline | 1368.1 (314.88) | 12212.2 (283.36)
  Week 26 | 1366.5 (316.94) | 979.8 (321.45)
  Overall percent change from Baseline to Week 26 | 1.3 (19.22) | -18.9 (19.44)

5. Secondary Outcome: Overall Change From Baseline to Week 26 in Child Health Assessment Questionnaire/Health Assessment Questionnaire (CHAQ/HAQ) Disability Index Score
Description: CHAQ/HAQ) = Patient questionnaire that measures the degree of disability on a scale of 0 (no disability) to 3 (maximal disability). A lower score indicates a greater response.
Time Frame: Baseline to week 26
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Aldurazyme Treatment
Number analyzed (Participants) | 23 | 21
Units on a scale
  Baseline | 1.9 (0.60) | 2.0 (0.49)
  Week 26 | 1.8 (0.71) | 1.9 (0.58)
  Overall change from Baseline to Week 26 | -0.1 (0.43) | -0.2 (0.39)

6. Secondary Outcome: Overall Change From Baseline to Week 26 in Active Joint Range of Motion (ROM)
Description: Active Joint Range of Motion (ROM): Shoulder Flexion Ability to maximally raise one's arm overhead without assistance. Shoulder range of motion (mean of left and right arms) measured in degrees (0-180) by goniometry. Greater degree of flexion indicates greater response.
Time Frame: Baseline to Week 26
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Placebo | Aldurazyme Treatment
Number analyzed (Participants) | 23 | 19
Degrees
  Baseline | 89.8 (23.99) | 96.1 (30.25)
  Week 26 | 85.2 (32.66) | 88.9 (37.69)
  Overall change from baseline to week 26 | -4.6 (27.18) | -1.2 (29.78)

7. Secondary Outcome: Overall Percent Change From Baseline to Week 26 in Urinary Glycosaminoglycan (GAG) Levels
Description: Urinary Glycosaminoglycan (GAG) Levels: Concentration of GAG relative to creatinine in urine. A greater decrease in GAG level indicates a greater response.
Time Frame: Baseline to Week 26
Measure: Mean (Standard Deviation); unit: ug/mg
Arm/Group | Placebo | Aldurazyme Treatment
Number analyzed (Participants) | 22 | 21
ug/mg
  Baseline | 183.3 (72.05) | 188.9 (60.93)
  Week 26 | 250.2 (105.09) | 81.3 (26.36)
  Overall Percentage of Change in GAG Level | 47.3 (59.34) | -54.1 (19.49)

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Groups:
- Placebo***Check Title***: Placebo***Check Description***
- Aldurazyme***Check Title***: Aldurazyme***Check Description***
Arm/Group | Placebo***Check Title*** | Aldurazyme***Check Title***
Serious Adverse Events (participants affected / at risk) | 0/23 | 3/22
Other Adverse Events (participants affected / at risk) | 23/23 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo***Check Title*** (N=23) | Aldurazyme***Check Title*** (N=22)
Cardiac arrest (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Ventriculoperitoneal shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo***Check Title*** (N=23) | Aldurazyme***Check Title*** (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2
Lymphatic disorder (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 8 | 1
Blepharitis (Eye disorders) | 1 | 0
Corneal opacity (Eye disorders) | 0 | 2
Eye discharge (Eye disorders) | 1 | 2
Eye pain (Eye disorders) | 0 | 1
Eye swelling (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dental discomfort (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 7
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 1
Tooth discolouration (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 9 | 5
Application site rash (General disorders) | 0 | 1
Catheter site related reaction (General disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 2 | 1
Face oedema (General disorders) | 0 | 2
Facial pain (General disorders) | 2 | 0
Fatigue (General disorders) | 4 | 1
Feeling hot (General disorders) | 1 | 2
Gait disturbance (General disorders) | 2 | 0
Gravitational oedema (General disorders) | 0 | 2
Hernia pain (General disorders) | 1 | 0
Influenza like illness (General disorders) | 3 | 0
Infusion site swelling (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 2
Injection site reaction (General disorders) | 2 | 4
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 13 | 8
Hepatomegaly (Hepatobiliary disorders) | 6 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Corneal graft rejection (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 2 | 0
Abscess (Infections and infestations) | 0 | 2
Catheter site infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 4 | 3
Fungal infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lice infestation (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 8 | 4
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 3 | 0
Otitis media chronic (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Sputum purulent (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 7
Urinary tract infection (Infections and infestations) | 3 | 2
Viral infection (Infections and infestations) | 2 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Bacteria urine (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 2 | 3
Brain scan abnormal (Investigations) | 0 | 1
Breath sounds abnormal (Investigations) | 4 | 2
Cardiac murmur (Investigations) | 3 | 2
Gallop rhythm present (Investigations) | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Nitrite urine present (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint crepitation (Musculoskeletal and connective tissue disorders) | 2 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 4 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 16 | 11
Hyperaesthesia (Nervous system disorders) | 1 | 0
Hyperreflexia (Nervous system disorders) | 0 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 3
Sinus headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0
Menstrual discomfort (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 8
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin swelling (Skin and subcutaneous tissue disorders) | 1 | 0
Ear tube removal (Surgical and medical procedures) | 1 | 0
Flushing (Vascular disorders) | 4 | 5
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Poor venous access (Vascular disorders) | 0 | 3

LIMITATIONS AND CAVEATS:
Rare disease with limited sample size, FVC calculations less reliable for patients whose height is below the 3rd% for general population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.